CLINICAL TRIAL: NCT01412398
Title: Special Drug Use Investigation of Fosrenol (Investigation for Patients With Continuous Ambulatory Peritoneal Dialysis)
Brief Title: Fosrenol Post-marketing Surveillance for Continuous Cyclic Peritoneal Dialysis in Japan
Acronym: FOSRENOL-CAPD
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15076
Record Dates: First submitted 2011-08-04; First posted 2011-08-09 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Hyperphosphatemia
Keywords: Fosrenol; Hyperphosphatemia; Continuous Cyclic Peritoneal Dialysis
MeSH Terms: conditions — Hyperphosphatemia | interventions — lanthanum carbonate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Drug (incl. Placebo)
  Interventions: Drug: Lanthanum Carbonate (Fosrenol, BAY77-1931) - chewable tablet

INTERVENTIONS:
Drug: Lanthanum Carbonate (Fosrenol, BAY77-1931) - chewable tablet — Patients in CAPD who have received Fosrenol for hyperphosphatemia

SUMMARY:
This study is a regulatory post marketing surveillance in Japan, and it is a local prospective and observational study of patients in continuous ambulatory peritoneal dialysis (CAPD) who have received Fosrenol for hyperphosphatemia. The objective of this study is to assess safety and efficacy of using Fosrenol in clinical practice. This study is also all case investigation of which the enrollment period is one year, and all patients in CAPD who received Fosrenol for hyperphosphatemia will be recruited and followed one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing continuous ambulatory peritoneal dialysis who received Fosrenol for hyperphosphatemia

Exclusion Criteria:

* Patients who are contraindicated based on the product label

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is all case investigation of which the enrollment period is one year, and all patients in CAPD who received Fosrenol for hyperphosphatemia will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2009-04-07 (Actual); Primary Completion 2014-04-08 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions in subjects who received Fosrenol | After Fosrenol administration, up to 1 year
Incidence of serious adverse events in subjects who received Fosrenol | After Fosrenol administration, up to 1 year

SECONDARY OUTCOMES:
Incidence of adverse drug reactions in subpopulation with baseline data [such as demographic data, concomitant disease, duration of treatment, maximum daily dose] and dose of Fosrenol | After Fosrenol administration, up to 1 year
Effectiveness evaluation assessment [achievement rate of a goal phosphate level; 3.5-6 mg/dL] | After Fosrenol administration, up to 1 year
Effectiveness evaluation assessment [achievement rate of a goal calcium level; 8.4-10.0 mg/dL] | After Fosrenol administration, up to 1 year
Clinical test value collections [calciotropic hormones, bone turnover markers] | After Fosrenol administration, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan